CLINICAL TRIAL: NCT05918094
Title: Comparing Modified XELOX Plus Sintilimab With Standard XELOX Plus Sintilimab in First-line Treatment for HER2-negative Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Rui-hua Xu, MD, PhD, Professor, President, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: mXELOX SYSUCC
Record Dates: First submitted 2023-06-15; First posted 2023-06-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; anti-PD-1; modified chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: 540 subjects will be randomized in a 1:1 ratio into either the modified XELOX plus sintilimab group or the standard XELOX plus sintilimab group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified XELOX + sintilimab (Experimental): The treatment option for the modified XELOX group (study group) is 200 mg of sintilimab IV Drip Q3W, 600 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 78 mg/m2 IV Drip Q3W. After 6 cycles of treatment, patients could choose capecitabine + sintilimab maintenance with a maximum treatment duration of 2 years.
  Interventions: Drug: Experimental dose: modified XELOX + sintilimab
- Standard XELOX + sintilimab (Active Comparator): The treatment option for the standard XELOX group (control group) is 200 mg of sintilimab IV Drip Q3W, 1000 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 130 mg/m2 IV Drip Q3W. After 6 cycles of treatment, patients could choose capecitabine + sintilimab maintenance with a maximum treatment duration of 2 years.
  Interventions: Drug: Standard dose: standard XELOX + sintilimab

INTERVENTIONS:
Drug: Experimental dose: modified XELOX + sintilimab — The treatment option for the modified XELOX group (study group) is 200 mg of sintilimab IV Drip Q3W, 600 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 78 mg/m2 IV Drip Q3W.
  Arms: Modified XELOX + sintilimab
Drug: Standard dose: standard XELOX + sintilimab — The treatment option for the standard XELOX group (control group) is 200 mg of sintilimab IV Drip Q3W, 1000 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 130 mg/m2 IV Drip Q3W.
  Arms: Standard XELOX + sintilimab

SUMMARY:
This is a randomized, controlled, multicenter phase Ⅲ study to evaluate the therapeutic efficacy of modified XELOX plus sintilimab versus standard XELOX plus sintilimab in subjects with advanced HER2-negative gastric or gastroesophageal adenocarcinoma in the first-line treatment. The primary outcome is the progression-free survival (PFS), with a planned enrollment of 540 subjects.

DETAILED DESCRIPTION:
Subjects will be randomized in a 1:1 ratio into either the modified XELOX plus sintilimab group or the standard XELOX plus sintilimab group. The treatment option for the modified XELOX group (study group) is 200 mg of sintilimab IV Drip Q3W, 600 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 78 mg/m2 IV Drip Q3W. The treatment option for the standard XELOX group (control group) is 200 mg of sintilimab IV Drip Q3W, 1000 mg/m2 of capecitabine PO BID for day 1-14, and oxaliplatin 130 mg/m2 IV Drip Q3W. After 6 cycles of treatment, patients could choose capecitabine + sintilimab maintenance with a maximum treatment duration of 2 years.

The primary endpoint of this study is the progression-free survival (PFS), defined as the time from random assignment of the subject to disease progression or death from any cause.

All eligible patients will be randomly assigned to either the trial or control group in a 1:1 ratio based on the following stratification factors: Whether the PD-L1 CPS score >= 5; Whether the age >70 years old.

ELIGIBILITY:
Inclusion Criteria:

* Have a good understanding of the study, are willing to follow the requirements of the study, and voluntarily sign the informed consent form.
* Aged ≥ 18 years old and ≤ 75 years old.
* Locally advanced unresectable or metastatic gastric or gastroesophageal adenocarcinoma confirmed by pathological histology or cytology.
* No previous systemic therapy. Note: Patients who have previously received neoadjuvant or adjuvant therapy may be enrolled if they have ended treatment without recurrence or disease progression for at least 6 months.
* Agree to provide a previously stored tumor tissue sample or a biopsy to collect tumor tissue.
* ECOG PS score is in the range of 0~1.
* Expected survival time ≥ 3 months.
* Subjects having adequate organ and bone marrow functions with laboratory test values within 7 days prior to enrollment meeting the following requirements (no blood components, cell growth factors, albumin, and other corrective therapy drugs are allowed to be given within the first 14 days of obtaining laboratory tests), as follows:

  1. Blood routine: absolute neutrophil count (ANC) ≥ 1.5×10^9/L; platelet count (PLT) ≥ 75×10^9/L; hemoglobin level (HGB) ≥ 7.5 g/dL.
  2. Liver function: serum total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN in subjects without liver metastases, and ALT and AST ≤ 5.0 × ULN in subjects with liver metastases; serum albumin ≥ 25 g/L.
  3. Renal function: serum creatinine (Cr) ≤ 1.5 x ULN, or creatinine clearance>50 mL/min.
* Female subjects of childbearing age or male subjects whose sexual partners are at childbearing age are required to take effective contraception measures throughout the treatment period and for 6 months after the treatment

Exclusion Criteria:

* Prior exposure to any immune checkpoint inhibitors (anti-PD-1 antibody, anti-PD-L1 antibody, CTLA-4 antibody).
* Receiving antitumor cytotoxic drugs, biological drugs (such as monoclonal antibodies), immunotherapy (such as interleukin 2 or interferon), or other investigational treatments within 4 weeks prior to enrollment.
* Receiving radiotherapy within 4 weeks prior to the first dose.
* Have undergone major surgical surgery within 4 weeks prior to enrollment or have not fully recovered from previous surgery.
* Known presence of symptomatic CNS metastases and/or carcinomatous meningitis. Subjects with prior treatment for brain metastases may participate in the study provided that the brain metastases have remained stable for at least 4 weeks prior to the first dose of study treatment; and that neurological symptoms have recovered to ≤ grade 1 by NCI CTCAE version 5.0.
* A history of other primary malignancies, except: malignancies in complete response for at least 2 years prior to enrollment and requiring no other treatment during the study period; adequately treated non-melanoma skin cancer or malignant freckled nevus with no evidence of disease recurrence; adequately treated carcinoma in situ with no evidence of disease recurrence.
* Active autoimmune disease requiring systemic therapy (e.g., use of disease-relieving drugs, corticosteroids, or immunosuppressants) within 2 years prior to the first dose. Alternative therapies (e.g., thyroxine, insulin, or physiologic corticosteroids for adrenal or pituitary insufficiency) are allowed. A known history of primary immunodeficiency. For patients with only positive autoimmune antibodies, the presence of autoimmune diseases should be confirmed at the discretion of the investigator.
* A history of gastrointestinal perforation and/or fistula in the previous 6 months.
* Presence of intestinal obstruction (including incomplete intestinal obstruction requiring parenteral nutrition).
* Confirmed as HER2-positive (i.e., IHC 3+ or IHC 2+ with ISH+) gastric or gastroesophageal adenocarcinoma.
* Have heart symptoms or diseases that are not well controlled, such as:

  1. Have had NYHA grade 3 or 4 cardiac insufficiency within 6 months prior to enrollment;
  2. Unstable angina;
  3. Have had acute myocardial infarction within 6 months prior to enrollment;
  4. Have had clinically significant arrhythmias within 6 months prior to enrollment requiring treatment or intervention.
* Infected with human immunodeficiency virus (HIV) (HIV 1/2 antibody or HIV RNA positive).
* Known to have acute or chronic active hepatitis B (HBsAg positive and HBV DNA ≥ 1000 copies/mL) or acute or chronic active hepatitis C (HCV antibody positive and HCV RNA positive).
* Severe infections that are in the active phase or poorly controlled in clinical practice. Serious infection, including but not limited to hospitalization for complications of infection, bacteremia or severe pneumonia, within 4 weeks prior to the first dose.
* A known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
* A history of allergy or known intolerance to any drug in the study regimen.
* Receiving live attenuated vaccine within 4 weeks prior to the first dose or planning to receive during the study period.
* The toxicity of previous antitumor therapy has not returned to grade 0-1 according to CTCAE 5.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 540 (Estimated)
Dates: Start 2023-04-30 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | an average of 4 years
  Time from randomization to disease progression or death from any cause

SECONDARY OUTCOMES:
Objective Response Rates (ORR) | an average of 4 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR) or partial response (PR) according to RECIST 1.1.
Overall Survival (OS) | an average of 4 years
  Time from randomization to death from any cause
Disease Control Rate (DCR) | an average of 4 years
  The percentage of subjects whose therapeutic effect evaluation is complete response (CR), partial response (PR) or stable disease (SD) according to RECIST 1.1.
Duration of Response (DOR) | an average of 4 years
  Time from achievement of a response to disease progression.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-C30 (EORTC QLQ-C30) | an average of 4 years
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit. The higher score means the worse quality of life.
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-STO22 (EORTC QLQ- STO22) | an average of 4 years
  Quality of life in patients with colorectal cancer is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) STO22. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit. The higher score means the worse quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, MD, Principal Investigator — Sun Yat-sen University
Locations (10):
- China (10):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The Affliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Tongji Hospital Affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No